CLINICAL TRIAL: NCT06240962
Title: Effects of Mindfulness Practice With Strength Training on Pain, Kinesiophobia and Function Among Sprinters With Patellofemoral Syndrome
Brief Title: Mindfulness Practice vs Strength Training on Pain, Kinesiophobia and Function Among Sprinters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0434
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Resistance Training; Patellofemoral Pain Syndrome; Kinesiophobia; Sprinters
Keywords: Mindfulness Practice; Resistance Training; Pain; Sprinters; Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Kinesiophobia; Pain | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training (Other): They will receive the strength training only will follow a protocol (6 weeks, 3 sessions/week) that feature training modifications to help control injury-related symptoms.
  Interventions: Other: Strength Training
- Mindfulness Exercise (Other): They will receive the mindfulness-exercise group will receive an 6-week mindfulness intervention in addition to the strength training protocol.
  Interventions: Other: Mindfulness Exercise

INTERVENTIONS:
Other: Strength Training — They will receive the strength training only (6 weeks, 3 sessions/week) that feature training modifications to help control injury-related symptoms.
  Arms: Strength Training
Other: Mindfulness Exercise — They will receive mindfulness-exercise for 6-week mindfulness intervention in addition to the strength training protocol.
  Arms: Mindfulness Exercise

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive the strength training only. Group B will receive the mindfulness-exercise in addition to the strength training protocol.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of mindfulness practice with strength training on pain, kinesiophobia and function among sprinters with patellofemoral syndrome. The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive the strength training only. Group B will receive the mindfulness-exercise in addition to the strength training protocol. Usual pain, pain during stepping, and pain during running will be assessed using visual analog scales. Functional limitations of the knee will be assessed using the Knee Outcome Survey. Fear of movement, pain catastrophizing, and coping strategies will be measured via the Tampa Scale for Kinesiophobia, the Pain Catastrophizing Scale, and the Coping Strategies Questionnaire, respectively. For strength training we will use Muscle-strengthening Exercise Questionnaire Short Form (MSEQ). These outcomes will be assessed at baseline and after 6 weeks

The data will be analyzed by SPSS, version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Males and Female between the ages of 18 and 40 years, Report running ≥2 times per week for >45 minutes or a minimum weekly running distance of 10 km, Present a history of insidious onset of signs and symptoms of PFP in 1 or both knees that was unrelated to trauma for at least 3 months before assessment, score <85/100 on the Activities of Daily Living Scale and Sports related of the Knee Outcome Survey (KOS-ADLS)

Exclusion Criteria:

* Intra-articular condition, Coexisting lower limb injury, History of patellar dislocation or knee surgery, Osgood-Schlatter or Sinding- Larsen-Johansson syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Knee Pain | pre and 6 weeks post interventional
  Usual pain, pain during stepping and running will be assessed using visual analog scales.
Kinesiophobia | pre and 6 weeks post interventional
  Tampa Scale will be used to assess kinesiophobia.
Physical Function | pre and 6 weeks post interventional
  Functional limitations of the knee will be assessed using the Knee Outcome Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Malik, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopes AD, Hespanhol Junior LC, Yeung SS, Costa LO. What are the main running-related musculoskeletal injuries? A Systematic Review. Sports Med. 2012 Oct 1;42(10):891-905. doi: 10.1007/BF03262301. PMID 22827721
- [Background] Witvrouw E, Callaghan MJ, Stefanik JJ, Noehren B, Bazett-Jones DM, Willson JD, Earl-Boehm JE, Davis IS, Powers CM, McConnell J, Crossley KM. Patellofemoral pain: consensus statement from the 3rd International Patellofemoral Pain Research Retreat held in Vancouver, September 2013. Br J Sports Med. 2014 Mar;48(6):411-4. doi: 10.1136/bjsports-2014-093450. No abstract available. PMID 24569145
- [Background] Domenech J, Sanchis-Alfonso V, Espejo B. Changes in catastrophizing and kinesiophobia are predictive of changes in disability and pain after treatment in patients with anterior knee pain. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2295-300. doi: 10.1007/s00167-014-2968-7. Epub 2014 Apr 2. PMID 24691626
- [Background] Mansfield CB, Selhorst M. The effects of fear-avoidance beliefs on anterior knee pain and physical therapy visit count for young individuals: A retrospective study. Phys Ther Sport. 2018 Nov;34:187-191. doi: 10.1016/j.ptsp.2018.10.008. Epub 2018 Oct 18. PMID 30368045
- [Background] Domenech J, Sanchis-Alfonso V, Lopez L, Espejo B. Influence of kinesiophobia and catastrophizing on pain and disability in anterior knee pain patients. Knee Surg Sports Traumatol Arthrosc. 2013 Jul;21(7):1562-8. doi: 10.1007/s00167-012-2238-5. Epub 2012 Oct 19. PMID 23081711
- [Background] Smith BE, Moffatt F, Hendrick P, Bateman M, Rathleff MS, Selfe J, Smith TO, Logan P. The experience of living with patellofemoral pain-loss, confusion and fear-avoidance: a UK qualitative study. BMJ Open. 2018 Jan 23;8(1):e018624. doi: 10.1136/bmjopen-2017-018624. PMID 29362256
- [Background] Piva SR, Fitzgerald GK, Wisniewski S, Delitto A. Predictors of pain and function outcome after rehabilitation in patients with patellofemoral pain syndrome. J Rehabil Med. 2009 Jul;41(8):604-12. doi: 10.2340/16501977-0372. PMID 19565153
- [Background] Rathleff MS, Rasmussen S, Olesen JL. [Unsatisfactory long-term prognosis of conservative treatment of patellofemoral pain syndrome]. Ugeskr Laeger. 2012 Apr 9;174(15):1008-13. Danish. PMID 22487407